CLINICAL TRIAL: NCT06481904
Title: An Observational, Long-term Safety Study of TZIELD® (Teplizumab-mzwv) in Patients With Stage 2 Type 1 Diabetes
Brief Title: Registry for Stage 2 Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18117; U1111-1306-6690 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- TZIELD group: Patients prior to the initiation of TZIELD treatment or initiated TZIELD treatment within 6 months to study enrollment
  Interventions: Drug: TZIELD (teplizumab-mzwv)
- Comparator group: Patients not planned to be treated

INTERVENTIONS:
Drug: TZIELD (teplizumab-mzwv) — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.
  Groups: TZIELD group

SUMMARY:
Stage 2 Type 1 Diabates (T1D) is an early stage of T1D characterized by dysglycemia but not yet leading to clinical symptoms. Progression of the disease to Stage 3 (clinical T1D), leads to overt hyperglycemia requiring eventually exogenous insulin.

TZIELD® (teplizumab-mzwv) has been approved to delay onset of stage 3 T1D, by the United States (US) Food and Drug Administration (FDA) for adults and children aged 8 years and older with Stage 2 T1D.

The purpose of this study is to collect general information on patients with stage 2 T1D and further information on the long-term effects of TZIELD® in patients with Stage 2 T1D, treated as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

TZIELD-Exposed Cohort

* Patients in the US diagnosed with Stage 2 T1D who are planned to initiate TZIELD treatment according to the currently approved label or who have initiated TZIELD treatment within 6 months prior to enrollment:
* Day 1: 65 mcg/m2
* Day 2: 125 mcg/m2
* Day 3: 250 mcg/m2
* Day 4: 500 mcg/m2
* Days 5 through 14: 1,030 mcg/m2 per day
* Cumulative dose is approximately 11,240 mcg/m2
* Appropriate written informed consent/assent as applicable for the age of the patient

TZIELD-Unexposed Cohort

* Patients in the US diagnosed with Stage 2 T1D but who are not treated with TZIELD
* Appropriate written informed consent/assent as applicable for the age of the patient

Exclusion Criteria:

* Patients who initiated TZIELD treatment more than 6 months prior to enrollment
* Patients who had participated in a previous clinical trial for TZIELD
* Patients in an ongoing clinical trial of an investigational product or who had ended participation within 6 months prior to study enrollment; patients participating in other observational studies may be enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the US diagnosed with Stage 2 Type 1 Diabetes
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2037-01-15 (Estimated); Study Completion 2037-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events of special interests (AESI) | Throughout the study, approximately 10 years
  Presence of AESIs including cytokine release syndrome (CRS), serious infections, hypersensitivity reactions, lymphoproliferative disorders, and malignancies
Number of serious adverse events (SAE) | Throughout the study, approximately 10 years
Number of adverse events (AE) in mothers, fetuses, and infants exposed to TZIELD during pregnancy | From start of pregnancy to 12 months post-partum
Number of maternal pregnancy-related events | From start of pregnancy to 12 months post-partum
Developmental outcomes of the infant | From birth of infant to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (31):
- United States (31):
  - University of California Los Angeles Health- Site Number : 8400020, Los Angeles, California
  - University of California San Francisco - Mission Bay- Site Number : 8400005, San Francisco, California
  - University of Colorado Hospital- Site Number : 8400026, Aurora, Colorado
  - Yale University School of Medicine- Site Number : 8400025, New Haven, Connecticut
  - Nemours Children's Speciality Care- Jacksonville- Site Number : 8400006, Jacksonville, Florida
  - University of Chicago Medical Center- Site Number : 8400017, Chicago, Illinois
  - Riley Hospital for Children at IU Health- Site Number : 8400004, Indianapolis, Indiana
  - Norton Healthcare- Site Number : 8400030, Louisville, Kentucky
  - Johns Hopkins School of Medicine- Site Number : 8400031, Baltimore, Maryland
  - University of Michigan Health System - Ann Arbor- Site Number : 8400028, Ann Arbor, Michigan
  - Associated Endocrinologists, PC- Site Number : 8400039, Farmington Hills, Michigan
  - Corewell Health- Site Number : 8400009, Grand Rapids, Michigan
  - Mayo Clinic- Site Number : 8400010, Rochester, Minnesota
  - Children's Mercy Adelle Hall Campus- Site Number : 8400014, Kansas City, Missouri
  - Women and Children's Hospital of Buffalo- Site Number : 8400018, Buffalo, New York
  - Feinstein Institute for Medical Research (Northwell)- Site Number : 8400016, Manhasset, New York
  - Ten's Medical PC- Site Number : 8400027, Staten Island, New York
  - SUNY Upstate Medical University - Syracuse- Site Number : 8400007, Syracuse, New York
  - UNC Children's Hospital- Site Number : 8400008, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400024, Cincinnati, Ohio
  - Rainbow Babies And Children's Hospital- Site Number : 8400011, Cleveland, Ohio
  - Columbus Regional Healthcare- Site Number : 8400013, Columbus, Ohio
  - The Ohio State University- Site Number : 8400032, Columbus, Ohio
  - Hospital of The University of Pennsylvania- Site Number : 8400021, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia- Site Number : 8400029, Philadelphia, Pennsylvania
  - AM Diabetes & Endocrinology Center- Site Number : 8400012, Bartlett, Tennessee
  - Vanderbilt University Medical Center- Site Number : 8400023, Nashville, Tennessee
  - University of Texas - Southwestern Medical Center- Site Number : 8400003, Dallas, Texas
  - Texas Children's Hospital- Site Number : 8400002, Houston, Texas
  - University of Utah Health Care- Site Number : 8400019, Salt Lake City, Utah
  - United BioSource Corporation- Site Number : 8400001, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org